CLINICAL TRIAL: NCT06291831
Title: A Retrospective Observational Non-Interventional Study (NIS) to Assess Patient Characteristics and Healthcare Resource Use (HRU) Among COVID-19 Patients With or Without Nirmatrelvir/Ritonavir (PAXLOVID™) Treatment in the Kingdom of Bahrain.
Brief Title: A Study to Learn About the Use of Paxlovid in Patients With COVID-19 in the Kingdom of Bahrain.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671050; NCT06291831 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-02-29; First posted 2024-03-04 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: COVID-19 patients; Paxlovid use; Bahrain
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients receiving Nirmatrelvir; Ritonavir (PAXLOVID): Adult COVID-19 patients' Healthcare Resource Utilization (HRU) within the 30-day period following nirmatrelvir, ritonavir prescription.
  Interventions: Drug: nirmatrelvir, ritonavir
- Controls: Adults COVID-19 patient HRU within 30 days period following nirmatrelvir/ritonavir prescription
  Interventions: Other: Controls

INTERVENTIONS:
Drug: nirmatrelvir, ritonavir — Patients receiving Nirmatrelvir; Ritonavir (PAXLOVID)
  Groups: Patients receiving Nirmatrelvir; Ritonavir (PAXLOVID)
Other: Controls — Patients who do not receive Nirmatrevir/ritonavir (Paxlovid)
  Groups: Controls

SUMMARY:
The purpose of this study is to collect information on the:

* general information of a group of people such as their age, sex
* clinical information of the patients such as any other illness before having COVID 19.
* the number of COVID-19 patients who meet and follow the most up to date World Health Organization (WHO) recommendations for medication to treat COVID-19 (such as version 14, published 10Nov2023) compared to Kingdom of Bahrain national recommendations
* adult COVID-19 patients' health care resource use and outcomes within the 28-day period In adult patients with COVID-19 who have been prescribed nirmatrelvir and ritonavir treatment.

This study will be conducted in the Kingdom of Bahrain. The study will capture information of the adult COVID-19 outpatients and inpatients who have been prescribed nirmatrelvir, ritonavir treatment and those not treated with nirmatrelvir, ritonavir.

This study will have about 3000 patients treated with Paxlovid™ therapy and 1000 were not. The study will involve collection of patient information from medical records. The information collected can be either from papers or from computers.

The study will include patient information of those who:

* had COVID-19 infection during the study period from 16 February 2022 to 30 November 2022.
* are 18 years of age or older. This study will help to inform decision-making on use of Paxlovid at the national level.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:Age 18 years and older Patients with a diagnosis of COVID-19 whose information can be extracted from the I-Seha database

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a retrospective observational cohort study of patients diagnosed with COVID-19 in the Kingdom of Bahrain. Treated patients are defined as those have been prescribed nirmatrelvir, ritonavir and managed in the outpatient setting (eg, receiving medical treatment without being admitted to a hospital for COVID-19) while control group is those not treated with nirmatrelvir, ritonavir. Data will be from the I-Seha electronic medical records and descriptive analyses will be conducted for these two cohorts and will compare healthcare resource use in patients treated with nirmatrelvir, ritonavir and those not treated with nirmatrelvir, ritonavir.
Sampling Method: Non-Probability Sample
Enrollment: 3011 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Gulf FZ, Busaiteen, Bahrain

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Murad MM, Atkin SL, Wasif PW, Behzad AA, Husain AMJA, d'Hellencourt FL, Joury J, Aziz MA, Haridy H, Spinardi J, Wang L, Boland F, Kyaw MH, Al-Qahtani M. A Retrospective Observational Study on COVID-19 Patients Receiving Treatment with Nirmatrelvir/Ritonavir (PAXLOVID). Pulm Ther. 2025 Dec;11(4):645-659. doi: 10.1007/s41030-025-00316-z. Epub 2025 Oct 6. PMID 41051660
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible participants diagnosed with corona virus disease 2019 (COVID-19) in the Kingdom of Bahrain who were offered Paxlovid (nirmatrelvir, ritonavir) treatment between 16 February 2022 to 30 November 2022 (9.5 months) was included in this retrospective observational study. Data was retrieved from Kingdom of Bahrain national health information system [(I-Seha electronic health records (EHR)].
Pre-assignment Details: Available retrospective data was evaluated per objectives of this study in 2 months of this study (study start date: 13-Mar-2024 to study completion date: 14-May-2024).
Groups:
- Treated With Paxlovid: Participants who were diagnosed with COVID-19 and accepted offer for treatment with Paxlovid (nirmatrelvir, ritonavir) treatment in real world setting. No intervention was administered under this study.
- Not Treated With Paxlovid: Participants who were diagnosed with COVID-19 and declined offer for treatment with Paxlovid (nirmatrelvir, ritonavir) treatment. This reporting arm served as control group.
Period: Overall Study
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Started | 2005 | 1006
Completed | 2005 | 1006
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid | Total
Number analyzed (Participants) | 2005 | 1006 | 3011
Age, Customized [Count of Participants; unit: Participants]
  Age: 12-17 Years | 2 | 0 | 2
  Age: 18-29 Years | 457 | 204 | 661
  Age: 30-49 Years | 453 | 208 | 661
  Age: 50-64 Years | 485 | 201 | 686
  Age: 65-74 Years | 459 | 189 | 648
  Age: Greater than equal to 75 Years | 149 | 204 | 353
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1,005 | 489 | 1494
  Male | 1000 | 517 | 1517
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Arab | 1,668 | 916 | 2584
  Ethnicity: Asian | 291 | 79 | 370
  Ethnicity: Black/African/Caribbean | 8 | 3 | 11
  Ethnicity: Mixed/Multiple Ethnic Groups | 16 | 3 | 19
  Ethnicity: Persian | 1 | 0 | 1
  Ethnicity: White | 21 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified Based on Education
Description: Baseline was defined as one year before the index date. Index date was Paxlovid prescription written date or dispense date; if neither of them were available, the COVID-19 diagnosis date was used as the index date.
Time Frame: Baseline; from available retrospective data evaluated during 2 months of this study
Population: I-Seha EHR was used to retrieve the data in this study for evaluation of its objectives. Education information required for this outcome measure was not available in I-Seha EHR. Hence, there was no data that could be analyzed for this outcome measure.
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants Classified Based on Employment Status
Description: as for outcome 1
Time Frame: Baseline; from available retrospective data evaluated during 2 months of this study
Population: I-Seha EHR was used to retrieve the data in this study for evaluation of its objectives. Employment status information required for this outcome measure was not available in I-Seha EHR. Hence, there was no data that could be analyzed for this outcome measure.
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Height
Description: as for outcome 1
Time Frame: Baseline; from available retrospective data evaluated during 2 months of this study
Population: I-Seha EHR was used to retrieve the data in this study for evaluation of its objectives. Height information required for this outcome measure was not available in I-Seha EHR. Hence, there was no data that could be analyzed for this outcome measure.
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Weight
Description: as for outcome 1
Time Frame: Baseline; from available retrospective data evaluated during 2 months of this study
Population: I-Seha EHR was used to retrieve the data in this study for evaluation of its objectives. Weight information required for this outcome measure was not available in I-Seha EHR. Hence, there was no data that could be analyzed for this outcome measure.
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Body Mass Index (BMI)
Description: as for outcome 1
Time Frame: Baseline; from available retrospective data evaluated during 2 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study. BMI was extracted from records and method how it was collected originally was not known.
Measure: Median (Inter-Quartile Range); unit: Kilogram over meter square (Kg/m^2)
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 2005 | 1006
Kilogram over meter square (Kg/m^2) | 29 [25 to 33] | 29 [25 to 34]

6. Primary Outcome: Number of Participants Classified Based on Smoking Status
Description: as for outcome 1
Time Frame: Baseline; from available retrospective data evaluated during 2 months of this study
Population: I-Seha EHR was used to retrieve the data in this study for evaluation of its objectives. Smoking status information required for this outcome measure was not available in I-Seha EHR. Hence, there was no data that could be analyzed for this outcome measure.
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Number of Participants With at Least 1 Pre-existing Comorbidities
Description: Pre-existing comorbidities included: asthma, emphysema, chronic obstructive pulmonary disease (COPD), hypertension, diabetes, obesity, cerebrovascular disease, neurological disease, chronic kidney disease, chronic liver disease, malignancy. Baseline was defined as one year before the index date. Index date was Paxlovid prescription written date or dispense date; if neither of them were available, the COVID-19 diagnosis date was used as the index date.
Time Frame: Baseline; from available retrospective data evaluated during 2 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 2005 | 1006
Participants | 1709 | 920

8. Primary Outcome: Number of Participants Who Took at Least 1 Concomitant Medications for Pre-existing Comorbidities
Description: as for outcome 1
Time Frame: Baseline; from available retrospective data evaluated during 2 months of this study
Population: I-Seha EHR was used to retrieve the data in this study for evaluation of its objectives. Concomitant medications for pre-existing comorbidities information required for this outcome measure was not available in I-Seha EHR. Hence, there was no data that could be analyzed for this outcome measure.
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Number of Participants Who Used Antibiotics
Time Frame: Up to 24 months following COVID-19 diagnosis; from available retrospective data evaluated during 2 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 2005 | 1006
Participants
  For any cause | 530 | 320
  For COVID-19 | 118 | 103

10. Secondary Outcome: Number of Participants With Hospitalization for Any Cause
Time Frame: Up to 24 months following COVID-19 diagnosis; from available retrospective data evaluated during 2 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 2005 | 1006
Participants | 137 | 123

11. Secondary Outcome: Number of Participants With Intensive Care Unit (ICU) Admission for Any Cause
Time Frame: Up to 24 months following COVID-19 diagnosis; from available retrospective data evaluated during 2 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 2005 | 1006
Participants | 3 | 1

12. Secondary Outcome: Number of Participants Classified According to Length of Stay (LOS) in ICU for Any Cause
Time Frame: Up to 24 months following COVID-19 diagnosis; from available retrospective data evaluated during 2 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 3 | 1
Participants
  3 Days | 0 | 1
  6 Days | 1 | 0
  Missing | 2 | 0

13. Secondary Outcome: Number of Participants With Yes/no Questionnaire on Outpatient Visits
Time Frame: Up to 24 months following COVID-19 diagnosis; from available retrospective data evaluated during 2 months of this study
Population: I-Seha EHR was used to retrieve the data in this study for evaluation of its objectives. Participants with yes/no questionnaire on outpatient visits information required for this outcome measure was not available in I-Seha EHR. Hence, there was no data that could be analyzed for this outcome measure.
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants With Emergency Room (ER) Visits for Any Cause
Time Frame: Up to 24 months following COVID-19 diagnosis; from available retrospective data evaluated during 2 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 2005 | 1006
Participants | 298 | 155

15. Secondary Outcome: Number of Participants With Supplemental Oxygen Usage
Time Frame: Up to 24 months following COVID-19 diagnosis; from available retrospective data evaluated during 2 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 2005 | 1006
Participants | 21 | 11

16. Secondary Outcome: Number of Participants With Vasopressor Use
Time Frame: Up to 24 months following COVID-19 diagnosis; from available retrospective data evaluated during 2 months of this study
Population: I-Seha EHR was used to retrieve the data in this study for evaluation of its objectives. Participants with vasopressor use information required for this outcome measure was not available in I-Seha EHR. Hence, there was no data that could be analyzed for this outcome measure.
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Participants Who Used Invasive Mechanical Ventilation (IMV)
Time Frame: Up to 24 months following COVID-19 diagnosis; from available retrospective data evaluated during 2 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
Number analyzed (Participants) | 2005 | 1006
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality for both the reporting groups: up to 24 months following COVID-19 diagnosis and adverse events only for "Treated with Paxlovid" group: at Day 5 post Paxlovid course completion; from available retrospective data evaluated during 2 months of this study
Description: Adverse events were passively reported only for those participants who were treated with Paxlovid. Adverse events were not monitored or assessed for participants not treated with Paxlovid. Adverse events were reported as per records from I-Seha EHR. There was no specific medical dictionary.
Groups:
- Treated With Paxlovid: Eligible participants who had COVID-19 and were treated with nirmatrelvir, ritonavir treatment (PAXLOVIDTM). Their data was studied retrospectively in this study.
Arm/Group | Treated With Paxlovid | Not Treated With Paxlovid
All-Cause Mortality (participants affected / at risk) | 0/2005 | 0/1006
Serious Adverse Events (participants affected / at risk) | 0/2005 | 0/0
Other Adverse Events (participants affected / at risk) | 1427/2005 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated With Paxlovid (N=2005) | Not Treated With Paxlovid (N=0)
Impaired sense of taste / Bitterness (General disorders) | 1214 | 0
Impaired sense of smell (General disorders) | 2 | 0
Stomach/Abdominal pain (General disorders) | 47 | 0
Diarrhea (General disorders) | 365 | 0
Nausea/Vomiting (General disorders) | 44 | 0
Muscle aches (General disorders) | 88 | 0
Headache (General disorders) | 15 | 0
Cough (General disorders) | 5 | 0
Tiredness/Fatigue (General disorders) | 4 | 0
Dizziness (General disorders) | 8 | 0
Itching (General disorders) | 7 | 0
Leg (General disorders) | 4 | 0
Skin rash (General disorders) | 3 | 0
Loss of appetite (General disorders) | 4 | 0
Chest Pain/Heaviness (General disorders) | 4 | 0
Neck/Back Pain (General disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT06291831/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT06291831/SAP_001.pdf